CLINICAL TRIAL: NCT05259423
Title: The Effects on Children and Parents of Educating Parents About Ways to Play With Babies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Michele Lobo, Associate Professor, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1858581-1
Record Dates: First submitted 2022-02-03; First posted 2022-02-28 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Infant Development; Developmental Delay
Keywords: Education; Parents; Infant; Motor Activity; Cognition; Infant development; language development; Infant health
MeSH Terms: conditions — Learning Disabilities; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to receive the Enriched Education Program (EEP) or the Typical Education Program (TEP).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will not be aware of their group assignment as all families will receive education about nine play activities. Sealed envelopes created prior to enrollment will conceal assignments (i.e., appropriate educational materials) and the next envelope for the correct block [Block 1: typical development (TD), low SES; Block 2: TD, mid-high SES; Block 3 developmental delay (DD), low SES; Block 4: DD, mid-high SES] will be handed to families by the blind assessor at in-person visits or emailed to virtual participants by a team member not engaged in the blind assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Typical Development, Enriched Education Program (Experimental): Parents of infants with typical development (i.e, not meeting the eligibility criteria for early intervention services in the state of Delaware) will receive enriched play activity education based on key ingredients evidenced to advance infant development.
  Interventions: Other: Enriched Education Program
- Typical Development, Typical Education Program (Active Comparator): Parents of infants with typical development (i.e, not meeting the eligibility criteria for early intervention services in the state of Delaware) will receive typical play education based on usual education found in commonly used websites, apps, and books.
  Interventions: Other: Typical Education Program
- Developmental Delay, Enriched Education Program (Experimental): Parents of infants with/at risk for developmental delay (i.e, meeting the eligibility criteria for early intervention services in the state of Delaware) will receive enriched play activity education based on key ingredients evidenced to advance infant development.
  Interventions: Other: Enriched Education Program
- Developmental Delay, Typical Education Program (Active Comparator): Parents of infants with/at risk for developmental delay (i.e, meeting the eligibility criteria for early intervention services in the state of Delaware) will receive typical play education based on usual education found in commonly used websites, apps, and books.
  Interventions: Other: Typical Education Program

INTERVENTIONS:
Other: Enriched Education Program — Enriched play activity education including 9 different activities each with 3 levels depending on the infant's current head and trunk control. Parents will be instructed to complete 3 activities each day for at least 5 minutes each for a total of 15 minutes per day.
  Arms: Developmental Delay, Enriched Education Program; Typical Development, Enriched Education Program
Other: Typical Education Program — Typical play activity education including 9 activities commonly described by popular parenting websites, mobile applications, and books. Parents will be instructed to complete 3 activities each day for at least 5 minutes each for a total of 15 minutes per day.
  Arms: Developmental Delay, Typical Education Program; Typical Development, Typical Education Program

SUMMARY:
The purpose of this study is to determine whether educating parents about how to play with infants affects infant development or caregiver characteristics.

The project will comparatively evaluate the effects of two different play education programs on infants' development and on caregiver characteristics in a sample of infants with typical development and a sample of infants with/at risk for developmental delay.

DETAILED DESCRIPTION:
Parents are the primary source of interaction for their infants; they determine their infants' daily experiences and provide opportunities for growth and learning that have cascading, longitudinal effects. Early experiences may be even more important for infants who are at risk of developmental delays. In the United States, one out of every six children ages 3-17 will be diagnosed with one or multiple developmental disabilities, and the prevalence is growing. While some children with developmental disabilities or delays benefit from early intervention (EI) services in this critical period, enrollment rates for eligible children are disturbingly low, with only 5-10% of children with delays receiving EI services at 24 months of age. For these children who do not receive EI services during this critical window for neuroplasticity and learning, parents are the primary persons tasked with independently creating opportunities for their infants' developmental growth. The purpose of this study is to improve our understanding of early parent education and to determine whether or how parent education changes child outcomes (i.e., developmental scores) and parental characteristics (i.e., physical and social setting, customs, parent psychology). The investigators will conduct a pilot randomized controlled trial with a parallel design enrolling parents and infants ages 1-6 months with typical development or with/at risk of developmental delays. The investigators will use blocked randomization to control for socioeconomic status, as this is a known factor that can impact infant development, to assign parent-infant dyads to receive either the Enriched Education Program (EEP) or the Typical Education Program (TEP). Parents will receive written, illustrated instructions describing nine play activities; they will be asked to perform three activities each day (5 minutes each, 15 minutes total per day), logging their activity for 4 weeks. EEP activities were designed to implement EI and developmental science principles, while TEP activities represent common activities described on parenting websites, books, and mobile applications. Participants will be evaluated longitudinally across five visits using a variety of measures of child development and parental characteristics: at pre-intervention (baseline), post-intervention (1 month), and at follow-up visits (1-, 2-, and 5-month follow-up). In addition, infants' motor milestone development will be tracked through the onset of walking. The effect of the interventions on child developmental outcomes and parental characteristics will be evaluated for infants with typical development and infants at risk/with developmental delays. Usability of the educational programs will also be evaluated. The results of this study may help inform future parent education interventions.

ELIGIBILITY:
Inclusion Criteria:

* Able to engage in the data collection activities and be available for either in-person or virtual visits
* Parent participating in the study must be at least 18 years of age
* Parent must be able to speak and read in English
* Parent must be physically capable of performing the play activities with their infant (i.e., able to carry the infant and play on the floor with the infant).
* If parents choose to participate virtually, they must report having a device with a camera and microphone for the use of Zoom and access to the internet.
* Infants must be between the ages of 1 month and 6 months at enrollment
* Infants must not be legally blind
* Infants who meet the criteria for the State of Delaware Early Intervention Inclusion Criteria will be included in the at-risk group. These criteria are: 1) established conditions, such as chromosomal disorders, genetic disorders, and neurologic disorders; or 2) developmental delay measured via a standardized developmental assessment (e.g., the DAY-C).

Exclusion Criteria:

* None beyond inclusion criteria

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Change in Infant Motor Development | Baseline (start of study), 1-month from start of study, 2-months from start of study, 3-months from start of study, 6-months from start of study
  Assessed with the Alberta Infant Motor Scale, an observational measure of motor performance in prone, supine, sitting, and standing positions through a total score and sub-scale scores. Total Score: Minimum: 0; Maximum: 60; Higher score indicating more advanced motor development
Change in Infant Developmental Outcomes | Baseline (start of study), 1-month from start of study, 2-months from start of study, 3-months from start of study, 6-months from start of study
  Assessed with the Developmental Assessment of Young Children- 2nd Edition, an assessment of motor, cognitive, and language development through subdomain and standard scores, as well as a general developmental index (normative cumulative score). Standard scores range from <70 to >130 with higher scores indicating more advanced development.
Change in Parental Play Behaviors: Positioning | Baseline (start of study), 1-month from start of study, 2-months from start of study, 3-months from start of study, 6-months from start of study
  A Naturalistic Play Assessment during which we can observe parents' typical daily interaction with infants (i.e., parents are asked to go about their typical activities as if the experimenter were not there) through behavioral coding play sessions lasting 10-20 minutes. We will video code information related to Positioning: Number of Bouts and percent time in prone, reclined, supine, side-lying, seated, standing, and held.
Change in Parental Play Behaviors: Handling | Baseline (start of study), 1-month from start of study, 2-months from start of study, 3-months from start of study, 6-months from start of study
  A Naturalistic Play Assessment during which we can observe parents' typical daily interaction with infants (i.e., parents are asked to go about their typical activities as if the experimenter were not there) through behavioral coding play sessions lasting 10-20 minutes. We will video code information related to Handling: Number of bouts and percent time with support by a container or parent at the head, upper trunk, lower trunk in prone, reclined, supine, side-lying, seated, standing, held positions.
Change in Parental Play Behaviors: Communication | Baseline (start of study), 1-month from start of study, 2-months from start of study, 3-months from start of study, 6-months from start of study
  A Naturalistic Play Assessment during which we can observe parents' typical daily interaction with infants (i.e., parents are asked to go about their typical activities as if the experimenter were not there) through behavioral coding play sessions lasting 10-20 minutes. We will video code information related to communication: Communication: Number of words (total and number unique), babbling, style (fluctuation in pitch, responsiveness/turn-taking, gestures while communicating, labeling objects).
Change in Parental Play Behaviors: Toys | Baseline (start of study), 1-month from start of study, 2-months from start of study, 3-months from start of study, 6-months from start of study
  A Naturalistic Play Assessment during which we can observe parents' typical daily interaction with infants (i.e., parents are asked to go about their typical activities as if the experimenter were not there) through behavioral coding play sessions lasting 10-20 minutes. We will video code information related to toys: Frequency of toy use, number of unique toys, location of toys (Number of bouts and percent time in reach; Number of bouts and Percent time within-grasp).
Usability and Feasibility of the Intervention | 1-month from start of study
  The usability and feasibility of both interventions (Enriched Education and Typical Education) will be assessed using a Perception Questionnaire with 7-point Likert Scales (1= Completely Disagree; 7 = Completely Agree) including the meaningfulness and ease of use of the activities.

SECONDARY OUTCOMES:
Change in Daily Positioning | 2 days surrounding each of the 5 visits: Baseline (start of study), 1-month from start of study, 2-months from start of study, 3-months from start of study, 6-months from start of study
  A position tracking garment, the get-around-garment will be worn during awake times for 2 days to determine the time spent in supine, prone, and upright positions.
Change in Infant Object Exploration | Baseline (start of study), 1-month from start of study, 2-months from start of study, 3-months from start of study, 6-months from start of study
  Assessed with the Object Exploration Assessment, which measures visual-manual interactions when infants are provided with specific objects (7) with varying properties for 30 seconds each to determine exploration time, bouts of exploration, individual behaviors (i.e., mouthing, looking, touching body, bilateral holding) and multimodal behaviors (i.e., looking while acting).
Change in Language Development | Baseline (start of study), 1-month from start of study, 2-months from start of study, 3-months from start of study, 6-months from start of study
  The Preschool Language Scales-5th Edition will be given to assess language development including preverbal, interaction-based language skills in the domains of auditory comprehension, and expressive communication standard scores as well as a total language score.
Change in Parental Beliefs about Development | Baseline (start of study), 1-month from start of study, 3-months from start of study, 6-months from start of study
  Parental beliefs will be measured with the Parental Beliefs on Motor Development scaled score and the Parental Knowledge and Beliefs Questionnaire which was developed to measure parent knowledge and beliefs about motor, cognitive and language development using 7-point Likert Scales. Items related to each developmental domain (motor, cognitive, language) will be summed to get a domain score in addition to a total score (sum).
Change in Parental Knowledge about Development | Baseline (start of study), 1-month from start of study, 3-months from start of study, 6-months from start of study
  Parental knowledge about language and cognitive development will be measured with the Survey of Parent/Provider Expectations and Knowledge and parent knowledge about motor development will be assessed with the Parental Knowledge and Beliefs Questionnaire using 7-point Likert Scales.Items related to each developmental domain (motor, cognitive, language) will be summed to get a domain score in addition to a total score (sum).
Change in Parent Beliefs and Knowledge about Play | Baseline (start of study), 1-month from start of study, 3-months from start of study, 6-months from start of study
  The Parent Play Questionnaire will survey parents' beliefs and knowledge about play with infants.
Change in Parenting Confidence | Baseline (start of study), 1-month from start of study, 3-months from start of study, 6-months from start of study
  The Karitane Parenting Confidence Scale will assess parents' confidence in their parenting abilities. Higher scores indicate greater parenting confidence.
Change in Parental Practices regarding Motor Development | Baseline (start of study), 3-months from start of study, 6-months from start of study
  The Motor Habits Questionnaire will be used to measure parents' practices regarding motor development.
Change in the Time of Achieving Developmental Milestones | Reported at Baseline (start of study) and reported at 1 month- intervals through the onset of independent walking (Typically 12 -15 months) or when the child reaches 24 months of age (whichever occurs first)
  The Parental Milestone Report will be used to track the timing of the development of key developmental milestones through the onset of independent walking.

OTHER OUTCOMES:
Affordances in the Home Environment Impact Child Developmental Outcomes and Parental Characteristics | Baseline (start of study)
  The Affordances in the Home Environment for Motor Development-Infant Scale will be used to survey the toys, space, and surfaces available in the home environment. Potential relationships between affordances in the home environment and child developmental outcomes and parental characteristics will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Michele A Lobo, PT, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Yes
A data sharing agreement is in place for the University of Delaware and the University of Chicago to share deidentified SPEAK-R and demographic data including: parent participant's age in years, highest level of school completed/highest degree obtained, race, and ethnicity age in years and highest level of school completed/highest degree obtained for other adult(s) living in the household, infant participant's race, ethnicity, and sex, and approximate total annual household income before taxes which the University of Chicago will use towards establishing the reliability of the SPEAK-R and publishing research articles.